CLINICAL TRIAL: NCT05539105
Title: A Prospective Observation Registry Study on the Alimentary Reconstruction After Radical Proximal Gastrectomy
Acronym: STAR-PG01
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STAR-PG01
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Proximal Gastric Adenocarcinoma; Reconstruction
Keywords: Proximal gastrectomy; Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Double tract reconstruction: Double tract reconstruction would be applied after proximal gastrectomy
  Interventions: Procedure: Double tract reconstruction
- Gastric conduit reconstruction: Gastric conduit reconstruction would be applied after proximal gastrectomy
  Interventions: Procedure: Gastric conduit reconstruction
- Other reconstructions: Other reconstructions except for double tract and gastric conduit reconstructions would be applied after proximal gastrectomy
  Interventions: Procedure: Other reconstructions

INTERVENTIONS:
Procedure: Double tract reconstruction — Double tract reconstruction would be applied after radical proximal gastrectomy.
  Groups: Double tract reconstruction
Procedure: Gastric conduit reconstruction — Gastric conduit reconstructionn would be applied after radical proximal gastrectomy.
  Groups: Gastric conduit reconstruction
Procedure: Other reconstructions — Other reconstructions except for double tract and gastric conduit reconstructions would be applied after radical proximal gastrectomy.
  Groups: Other reconstructions

SUMMARY:
This study is designed as a prospective, real world registry study that compare the safety and efficacy of the different construction methods after radical proximal gastrectomy.

DETAILED DESCRIPTION:
* The patient was admitted to the hospital, and at the time of physical examination, the following conditions were met: 18 years old ≤ age ≤ 80 years old; preoperative ECOG performance status score 0/1; non-pregnant or lactating women; no serious mental illness; no serious respiratory disease; No severe hepatic and renal insufficiency; no history of unstable angina pectoris and myocardial infarction within 6 months; no history of cerebral infarction or cerebral hemorrhage within 6 months, except for old cavity infarction; no history of continuous glucocorticoid therapy (local Except for applications); pulmonary function test showed FEV1 ≥ 50% of the predicted value. The patient did not participate in other clinical studies (within 6 months).

  * gastric adenocarcinoma was diagnosed by endoscopic examination and histopathological biopsy of the patient's primary lesion, including: papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly adherent carcinoma (including signet ring cell carcinoma and other types), Mixed adenocarcinoma, etc. In qualified units, endoscopic ultrasonography (EUS) is recommended. The tumor is located in the upper part of the stomach or at the esophagogastric junction (tumor diameter is less than 4cm, and the length of invasion of the esophagus is less than 2cm);

    * Enhanced CT scan of the abdomen and pelvis was performed on the patient. For upper gastric cancer, no tumor invading the muscular layer, subserosal layer or serosa layer was found, and no distant metastasis occurred; for esophagogastric junction cancer, no distant metastasis occurred;

      * The patient has a clear diagnosis of gastric adenocarcinoma, and it is expected that proximal gastrectomy and lymph node dissection can be performed to obtain an R0 surgical result. .

        * The patient's ASA is I-III. ⑥ At this point, the patient becomes a potential selected case and enters the case selection procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Tumor located in the upper or esophagogastric junction (EGJ), and curative resection with more than 1/2 remant is expected to be achievable by proximal gastrectomy with D2 lymphadenectomy (also apply to multiple primary cancers);
* Clinical stage T1NxM0 (According to AJCC-8th TNM staging system) of the upper stomach or diameter of EGJ cancer less than 4cm with invading esophgus no more than 2cm without any distant metastasis;
* Primary lesion is pathologically diagnosed as gastric adenocarcinoma, such as papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), and mixed adenocarcinoma;
* Preoperative performance status (ECOG，Eastern Cooperative Oncology Group) of 0 or 1
* Preoperative ASA (American Society of Anesthesiologists) scoring: I-III
* Sufficient organ functions
* Written informed consent

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, multi-center, open, observational, real-world registry study, prospectively and consecutively enrolling patients undergoing proximal gastric surgery in several important gastric cancer across the country. This study emphasizes the continuity of enrolled patients and the breadth of data sources to reflect the real clinical situation. This study plans to include about 10 centers across the country, and plans to enroll consecutive patients who will undergo radical proximal gastrectomy within 2 years. It is expected that a total of 600 prospective registry cases will be included.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflux esophagitis incidence 1 year after surgery | 1 year
  Reflux esophagitis refers to esophageal erosions and/or esophageal ulcers caused by the reflux of esophageal contents into the esophagus or above (oral mouth, throat, lungs) causing complaints of discomfort and endoscopic manifestations of esophageal mucosal defects.

SECONDARY OUTCOMES:
Morbidity after surgery | 30 days
  Take the total number of patients receiving surgical treatment as the denominator, and the number of patients with intraoperative/postoperative early and late complications during any one and follow-up as the numerator to calculate the proportion;
Body weight(kg) after surgery | 12 months
  Body weight(kg)would be monitored during follow-up after surgery.
Albumin(g/L) after surgery | 12 months
  Albumin(g/L) would be monitored during follow-up after surgery.
Hemoglobin(g/L) after surgery | 12 months
  Hemoglobin(g/L) would be monitored during follow-up after surgery.
3-year relapse free survival rate | 3 years
  The time between the date of surgery as the starting point and the date of tumor recurrence as the ending point (or the date of death due to tumor cause when the exact date of tumor recurrence is not known).
  When neither death nor tumor recurrence was observed at follow-up, the final date of confirmation of recurrence-free survival (final recurrence-free survival confirmation date: the last of the date of the outpatient visit or the date of the examination received) was used.
Mortality after surgery | 30 days
  Taking the total number of patients receiving surgical treatment as the denominator, and observing any of the following patients as the numerator, the ratio calculated as the surgical death ratio:
  1. According to the observation items during the operation and the observation items after the operation, it will be recorded as death;
  2. All patients who died from the start of the operation to within 30 days after the operation (including 30 days) (regardless of whether the cause of death was causally related to the operation);
  3. In a longer period of time after 31 days after the operation, there is definite evidence that the death of the patient has a direct causal relationship with the first operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided